CLINICAL TRIAL: NCT03061188
Title: Phase I/Ib Study of Nivolumab and Veliparib in Patients With Advanced Solid Tumors and Lymphoma With and Without Alterations in Selected DNA Repair Genes
Brief Title: Phase I/Ib Study of Nivolumab & Veliparib in Patients With Advanced Solid Tumors & Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); AbbVie (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Young Kwang Chae, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 16MH03; STU00204250 (Other: Northwestern University IRB); NU 16MH03 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-02018 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Neoplasm; Aggressive Non-Hodgkin Lymphoma; Recurrent Solid Neoplasm; Refractory Mantle Cell Lymphoma; T-Cell Non-Hodgkin Lymphoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — Nivolumab; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (veliparib, nivolumab) (Experimental): Patients receive veliparib PO BID on day 1 and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
The purpose of this research study is to determine the highest and safest dose of the experimental drug veliparib when combined with nivolumab. We will also study how safely this combination of medication can be given in advanced cancer and lymphoma and benefits of receiving this therapy. Nivolumab is currently approved in certain cancers such as melanoma, lung cancer and kidney cancer. Veliparib is not yet approved for use in the United States, and is considered experimental. Veliparib inhibits (blocks) the activity of the enzyme PARP. This blocking activity may prevent the cancer cell from repairing itself and resume growing. Nivolumab increases T cells in your immune system, which allows your immune system to attack the cancer. We think the combination of these drugs will be more effective against your cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify maximum tolerated dose (MTD) for the combination treatment of nivolumab and veliparib in patients with advanced refractory solid cancers and lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of nivolumab and veliparib in patients with advanced refractory solid cancers and lymphoma with and without mutations in selected DNA repair genes.

II. To evaluate the efficacy of treatment with nivolumab and veliparib in this population by objective response rate (ORR, defined as partial response [PR] + complete response [CR]), clinical benefit rate (CBR, defined as stable disease [SD] for >= 12 weeks, PR, + CR), and progression free survival (PFS, defined as the time from treatment initiation to documented disease progression) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria version (v)1.1 or Lugano criteria.

III. To evaluate efficacy of treatment with nivolumab and veliparib in this population by ORR, CBR, and immune-related PFS (irPFS) using irRECIST criteria.

IV. To evaluate overall survival (OS) in this population at 3 years from the start of treatment.

V. To evaluate the proportion of patients alive and progression free at 24 weeks in this population.

VI. To evaluate ORR to nivolumab and veliparib in patients with prior exposure to single agent PD-1/PD-L1 inhibitors.

TERTIARY OBJECTIVES:

I. To evaluate if any of the following predict response to veliparib in combination with nivolumab: tissue PD-L1 protein expression, immune cell infiltration markers.

II. To demonstrate the pharmacodynamic effects of veliparib and nivolumab on biomarkers including PD-L1, TILs, T cell subpopulations, and T cell receptor genotype.

III. To explore the pattern of clonal changes through circulating cell free DNA assay.

IV. To assess the dynamic change in both immune and genomic biomarkers in blood that may correlate with response to veliparib.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) twice daily (BID) on day 1 and nivolumab intravenously (IV) over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically documented (either primary or metastatic site) diagnosis of advanced solid tumor cancer (stage IV or unresectable) or aggressive lymphoma (diffuse large B cell lymphoma, mantle cell lymphoma, T cell lymphoma, and natural killer [NK] cell lymphoma)

  * NOTE: The following histologies will be excluded given known response to PD-1/PD-L1 inhibitor monotherapy: non-small cell lung cancer, squamous cell carcinoma of head and neck, melanoma, renal cell carcinoma, bladder cancer, Hodgkin's lymphoma, Merkel cell carcinoma, and high-frequency microsatellite instability (MSI-H) colorectal cancer
* All patients must have received, and be relapsed/refractory to at least one line of systemic therapy

  * NOTE: This does not include surgery or radiation alone; patients may have received any number of systemic therapies
* All patients with relapsed/refractory lymphoma must have received or be ineligible for autologous stem cell transplant or be ineligible for allogeneic stem cell transplant

  * NOTE: Patients must not have had a prior allogeneic stem cell transplant
* Patients must have measurable disease as per appropriate guidelines:

  * Solid tumors: by RECIST v1.1
  * Lymphoma: patient has at least one measurable nodal lesion (>= 2 cm) according to Lugano classification; if the patient has no measurable nodal lesions >= 2 cm in the long axis at screening, then the patient must have at least one measurable extra-nodal lesion
* Patients must have the ability to understand and the willingness to sign a written consent prior to registration in the study
* For expansion cohort patients, the profiling must reveal at least one mutation in the following selected DNA repair genes involved in cell cycle arrest signal transduction, BRCA1 pathway, Fanconi's proteins pathway, and RAD51 pathway: (ATR, ATM, CHEK1, CHEK2, BRCA1, BAP1, BARD1, FANCD2, FANCE, FANCC, RAD50, FANCA, RAD51, BRCA2, PALB2, CDK12 [ENSG00000167258, also known as CRK7, CRKR, CRKRS], POLE, POLD1, BRAC2, PRKDC, ERCC2, POLQ, MRE11A, NBN [MBS1]), or at least one gene amplification in FANCD2, FANCE, FANCC, FANCA, C11orf30 (EMSY)

  * NOTE: Tissue or blood cell free DNA are allowed for genomic profiling of tumor; profiling should have been performed at a Clinical Laboratory Improvement Act (CLIA) certified lab =< 1 year prior to registration
  * NOTE: Patients in the dose escalation phase are not required to have such mutations; although genomic profiling is not required for dose escalation patients, it is encouraged in these patients prior to or after study registration if feasible
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have adequate organ and bone marrow function =< 14 days prior to registration, as defined below (Note: blood transfusion or growth factors is not permitted within 14 days of registration):
* Absolute neutrophil count >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase and aspartate aminotransferase =< 5 x ULN
* Calculated creatinine clearance according to the Cockcroft and Gault equation >= 50 mL/min
* Females of child-bearing potential (FOCBP) and men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and the designated post-treatment period

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test =< 7 days prior to registration
* Patients must be able to swallow oral medication

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy =< 14 days prior to entering the study are not eligible

  * NOTE: Patients may not have had systemic chemotherapy within 28 days
* Patients are not eligible who have had major surgery =< 14 days of registration; please contact principle investigator (PI) and quality assurance monitor (QAM) for questions about specific surgical procedures
* Patients are not eligible who have received prior PARP inhibitors (including but not limited to veliparib, talazoparib, rucaparib, and olaparib)
* Patients are not eligible who have received systemic chemotherapy or investigational agents =< 28 days prior to registration
* Patients are not eligible who have received prior immunotherapy including interleukin-2 and immune checkpoint antagonists and/or agonists (including but not limited to PD-1, PD-L1, CD137, or OX40)

  * NOTE: Single agent anti-CTLA4 monoclonal antibody treatments are permitted; cancer vaccine therapies are permitted
* Patients with the following histologies are not eligible for either study cohort given known response to PD-1/PD-L1 inhibitor monotherapy:

  * Non-small cell lung cancer, squamous cell carcinoma of head and neck, melanoma, renal cell carcinoma, bladder cancer, Hodgkin's lymphoma, Merkel cell carcinoma, and MSI-H colorectal cancer
* Patients are not eligible who have had a prior allogeneic stem cell transplant

  * NOTE: Autologous stem cell transplant is acceptable
* Patients who are taking any herbal (alternative) medicines are NOT eligible for participation; patients must be off any such medications by the time of registration for >= 14 days

  * NOTE: Vitamin supplements are acceptable
* Patients must have no history of central nervous system (CNS) metastasis at the screening assessment

  * NOTE: Patients with stable brain metastases (mets) which have been treated are eligible; patients with suspected symptoms of CNS metastasis should undergo CNS imaging at the time of screening to rule out active metastasis
* Patients who have had a prior severe infusion reaction to a monoclonal antibody are not eligible
* Patients are not eligible who have a history of or active autoimmune disease within the past 3 years with the following exceptions:

  * Vitiligo or alopecia
  * Hypothyroidism on stable doses of thyroid replacement therapy
  * Psoriasis not requiring systemic therapy within the past 3 years
* Patients with a history of primary immunodeficiency disease or tuberculosis are not eligible
* Patients who have an uncontrolled current illness including, but not limited to any of the following, are not eligible:

  * Uncontrolled pulmonary, renal, or hepatic dysfunction
  * Ongoing or active infection requiring systemic treatment including hepatitis B and hepatitis C
  * Known active or chronic viral hepatitis or human immunodeficiency virus (HIV)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Clinically significant gastrointestinal disease or digestive dysfunction compromising absorption of veliparib
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients with a prior diagnosis of cancer must not have received treatment in the last 3 years prior to registration

  * NOTE: Patients with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* Patients must not have a history of prior stroke, transient ischemic attack (TIA), pulmonary embolism, or untreated deep vein thrombosis

  * NOTE: Patients may be eligible if they have received at least 3 months of anticoagulation for a deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young K. Chae, MD, MPH, MBA, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened for accrual on May 23, 2017 with goal of 50 patients. Due to funding issues the goal was reduced to 15. First patient started treatment June 1, 2017. Study design for Phase 1 was 3 + 3 escalation. The study closed Aug. 5, 2019 with accrual for the study design having been met.
Groups:
- Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab): Patients receive veliparib 200 mg (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab): Patients receive veliparib 300 mg (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab); Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab: Patients receive veliparib 400 mg (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
Period: Completed 1st Cycle
Arm/Group | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab
Started (The starting dose (Cohort 1) was not de-escalated.) | 0 | 3 | 6 | 6
Completed | 0 | 3 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Went on to Cycle 2 and Beyond
Arm/Group | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab
Started (The starting dose (Cohort 1) was not de-escalated.) | 0 | 3 | 6 | 6
Received Dose of Study Drugs | 0 | 3 | 5 | 5
Completed | 0 | 3 | 5 | 5
Not Completed | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Period: On Follow-up for 3 Years
Arm/Group | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab
Started (The starting dose (Cohort 1) was not de-escalated.) | 0 | 3 | 6 (Patients who received at least one dose of study drug go into follow-up.) | 6 (Patients who receive at least one dose of study drug go into follow-up.)
Completed | 0 | 0 | 1 | 1
Not Completed | 0 | 3 | 5 | 5
Not completed — Death | 0 | 3 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The starting dose (Cohort 1) was never de-escalated, so Cohort -1 never opened.
Groups:
- Velaparib PO Twice Daily + Nivolumab (Cohort -1): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose in Phase 1: Cohort -1: 200mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1)
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Velaparib PO Twice Daily + Nivolumab (Cohort 1): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose in Phase 1: Cohort 1: 300 mg,
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1)
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Velaparib PO Twice Daily + Nivolumab (Cohort 2): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose: 400 mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1)
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Velaparib PO Twice Daily + Nivolumab (Phase 2): Patients in all Phase 1 cohorts and Phase 2 receive velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose 400 mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1)
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Total: Total of all reporting groups
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort -1) | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2) | Velaparib PO Twice Daily + Nivolumab (Phase 2) | Total
Number analyzed (Participants) | 0 | 3 | 6 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 5 | 4 | 11
  >=65 years | 0 | 1 | 1 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 5 | 8
  Male | 0 | 3 | 3 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 3 | 6 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 3 | 5 | 4 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 6 | 6 | 15
Mutation in DNA repair gene present [Number; unit: participants] — Patients counted under "Yes" tested positive for a mutation in the following selected DNA repair genes (involved in cell cycle arrest signal transduction): BRCA1 pathway, Fanconi's proteins pathway, and RAD51 pathway: [ATR, ATM, CHEK1, CHEK2, BRCA1, BRIP1, BAP1, BARD1, FANCD2, FANCE, FANCC, RAD50, FANCA, RAD51, BRCA2, PALB2, CDK12 (ENSG00000167258, also known as CRK7, CRKR, CRKRS), POLE, POLD1, BRAC2, PRKDC, ERCC2, POLQ, MRE11A, NBN (MBS1)], or at least one gene amplification in FANCD2, FANCE, FANCC, FANCA, C11orf30 (EMSY).
  participants
    Yes |  | 1 | 3 | 5 | 9
    No |  | 2 | 3 | 1 | 6
Lymphoma vs Solid Tumor [Count of Participants; unit: Participants]
  Lymphoma | 0 | 0 | 0 | 0 | 0
  Solid Tumor | 0 | 3 | 6 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD will be defined as the highest dose that causes dose-limiting toxicities (DLTs) in <2 of 6 patients. Toxicity will be assessed using CTCAEv4.03. A DLT is defined as an Adverse Event (AE) or abnormal laboratory value assessed as at least possibly related to the study medication, occurs ≤ 28 days (1 cycle) following the first dose of veliparib and nivolumab and meets any of the following criteria:
  Grade ≥ 3 non-hematologic toxicities that represent at least a 2-grade increase from baseline excluding Nausea, vomiting, diarrhea lasting ≤48 hours, Electrolyte abnormalities resolving within ≤24 hours, Hypersensitivity reactions,and Alopecia.
  Grade 4 thrombocytopenia (platelets < 25.0 x 109 /L) Grade 3 thrombocytopenia with bleeding (platelets < 0.5 x 109 /L) 5. Grade 3 febrile neutropenia with fever lasting for > 7 days 6. Grade 4 febrile neutropenia of any duration 7. Dosing delay due to toxicity for > 14 consecutive days from the date nivolumab or veliparib is due.
Time Frame: First Cycle of Treatment with velaparib and nivolumab (28 days)
Measure: Number; unit: mg
Groups:
- Velaparib PO Twice Daily + Nivolumab (Phase 1): Patients in all Phase 1 cohorts receive velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  *Velaparib dose in Phase 1: Cohort -1: 200mg, Cohort 1: 300 mg, Cohort 2: 400 mg
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Phase 1)
Number analyzed (Participants) | 9
mg | 400

2. Secondary Outcome: Number of Participants With Adverse Events Possibly Related to Study Drugs Graded 3, 4, and 5
Description: Toxicity, both frequency and severity, will continue to be measured by monitoring the occurrence of adverse events. Adverse events will be defined as those included in CTCAE v 4.03. AEs that were determined to be at least possibly related to study drug and graded 3, 4, 5 are included here. Grade 1 (mild): the event causes discomfort without disruption of normal daily activities. Grade 2 (moderate): the event causes discomfort that affects normal daily activities. Grade 3 (severe): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status. Grade 4 (Life-threatening): the patient was at risk of death at the time of the event. Grade 5 (fatal): the event caused death.
Time Frame: Up to 30 days after treatment discontinuation, where 1 cycle =28 days, and range of cycles is 1-12.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab
Number analyzed (Participants) | 3 | 6 | 6
Participants
  Grade 3 Hypertension | 1 | 0 | 0
  Grade 3 Aspartate aminotransferase increased | 1 | 0 | 0
  Grade 3 Alanine aminotransferase increased | 1 | 0 | 0
  Grade 3 Alkaline phosphatase increased | 1 | 1 | 0
  Grade 3 Anemia | 1 | 2 | 0
  Grade 4 Anemia | 0 | 1 | 0
  Grade 3 Platelet count decreased | 0 | 1 | 0
  Grade 3 Fatigue | 0 | 2 | 0
  Grade 3 Hyponatremia | 0 | 1 | 0
  Grade 3 Hypokalemia | 0 | 1 | 0

3. Secondary Outcome: ORR (Overall Response Rate)
Description: Overall response rate or ORR, (partial response (PR) + complete response (CR)) will be evaluated using RECIST criteria v1.1 or Lugano 2014 classification for assessment of Lymphoma.
  Per RECIST v. 1.1: PR= : At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR= Disappearance of all target lesions.
  Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Per Lugano 2014 classification, scored on a Deauville 5-point scale (an internationally-recommended scale using FDG PET-CT in the initial staging and assessment of treatment response in Hodgkin lymphoma (HL) and certain types of non-Hodgkin lymphomas (NHL).
  * Partial metabolic response (PMR): score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size.
  * Complete metabolic response (CMR): Score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass
Time Frame: after 2 cycles at first response time point (1 cycle = 28 days)
Measure: Number; unit: participants
Groups:
- Velaparib PO Twice Daily + Nivolumab (Cohort 1): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose in Phase 1: Cohort 1: 300 mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1) Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV Pharmacological Study: Correlative studies Veliparib: Given PO
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2) | Velaparib PO Twice Daily + Nivolumab (Phase 2)
Number analyzed (Participants) | 3 | 6 | 6
participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR= stable disease for ≥12 weeks + Partial Response + Complete Response per RECIST v1.1 for solid tumors or Lugano 2014 classification for lymphomas. Lugano scored on a Deauville 5-point scale. RECIST v. 1.1: PR= : At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Lugano 2014 classification: PR: score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size. CR: Score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass. SD: No metabolic response, Score 4 or 5 with no significant change in FDG uptake from baseline at interim or end of treatment.
Time Frame: From the start of treatment and every 2 cycles during treatment where 1 cycle =28 days, average number of cycles is 4 and range of cycles is 1-12.
Measure: Number; unit: participants
Groups:
- Velaparib PO Twice Daily + Nivolumab (Cohort 1): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Velaparib dose in Phase 1: Cohort 1: 300 mg
  Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1) Laboratory
  Biomarker Analysis: Correlative studies
  Nivolumab: Given IV Pharmacological Study: Correlative studies
  Veliparib: Given PO
- Velaparib PO Twice Daily + Nivolumab (Phase 2): Patients in all Phase 1 cohorts and Phase 2 receive velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose 400 mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1) Laboratory Biomarker Analysis: Correlative studies Nivolumab: Given IV Pharmacological Study: Correlative studies Veliparib
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2) | Velaparib PO Twice Daily + Nivolumab (Phase 2)
Number analyzed (Participants) | 3 | 6 | 6
participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease for or ≥12 weeks | 0 | 4 | 2

5. Secondary Outcome: Progression Free Survival (PFS)
Description: To evaluate Progression Free Survival (PFS) for patients treated with nivolumab and veliparib, defined as the time from treatment initiation to documented disease progression. Evaluated by RECIST criteria v1.1 for solid tumors or Lugano 2014 classification for assessment of Lymphoma. RECIST v. 1.1 definition for PD (Progressive disease): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Lugano 2014 classification, scored on a Deauville 5-point scale (an internationally-recommended scale using FDG PET-CT in the initial staging and assessment of treatment response in Hodgkin lymphoma (HL) and certain types of non-Hodgkin lymphomas (NHL). Per Lugano criteria: Partial metabolic disease (PMD):Score 4 or 5 with an increase in intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
Time Frame: From the start of treatment and every 2 cycles during treatment, and up to three years, where 1 cycle =28 days, and range of cycles is 1-12.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Velaparib PO Twice Daily + Nivolumab (Cohort 2 + Phase 2): Velaparib (oral medication) twice daily and nivolumab IV over 30 minutes on days 1 and 15 of courses 1-4 and IV over 60 minutes on day 1 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Velaparib dose: 400 mg
  * Nivolumab dose: Cycle 1-4: 240 mg IV every 14 days (Days 1 & 15) + Cycle 5+: 480mg IV every 28 days (Day 1)
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Pharmacological Study: Correlative studies
  Veliparib: Given PO
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2 + Phase 2)
Number analyzed (Participants) | 3 | 11
months | 2.07 [2.00 to NA] — The upper limit of the confidence interval would be outside of the limits of the observed values and thus cannot be reported. | 1.94 [1.77 to NA] — The upper limit of the confidence interval would be outside of the limits of the observed values and thus cannot be reported.

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from treatment initiation until death due to any cause, assessed up to 3 years from the start of treatment.
Time Frame: From the start of treatment and up to 3 years, where 1 cycle =28 days, and range of cycles is 1-12.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2 + Phase 2)
Number analyzed (Participants) | 3 | 12
months | 5.82 [4.73 to NA] — 95% UCL for median survival was calculated by finding the smallest observed death time whose upper 95% CI was just above 0.5. but no observed death time met this criteria. | 11.79 [6.18 to NA] — 95% UCL for median survival was calculated by finding the smallest observed death time whose upper 95% CI was just above 0.5. but no observed death time met this criteria.

7. Secondary Outcome: Number of Patients Alive and Progression Free at 24 Weeks
Description: To evaluate the number of patients alive and progression free at 24 weeks. -Per RECIST v. 1.1 (for solid tumors) progression is defined as : At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.) -Lugano 2014 classification, scored on a Deauville 5-point scale (an internationally-recommended scale using FDG PET-CT in the initial staging and assessment of treatment response i Hodgkin lymphoma (HL) and certain types of non-Hodgkin lymphomas (NHL). Per Lugano criteria: Partial metabolic disease (PMD):Score 4 or 5 with an increase in intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment.
Time Frame: At 24 weeks
Population: 2 patients not included in these results as they came off treatment before 24 weeks - one withdrew consent and 1 came off treatment for palliative radiation.
Measure: Number; unit: participants
Arm/Group | Velaparib PO Twice Daily + Nivolumab (Cohort 1) | Velaparib PO Twice Daily + Nivolumab (Cohort 2) | Velaparib PO Twice Daily + Nivolumab (Phase 2)
Number analyzed (Participants) | 3 | 5 | 5
participants | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 3 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment, where 1 Cycle = 28 days the range of cycles attempted was 1-12.
Description: The starting dose was Cohort level 1. There were no dose-limiting toxicities on Cohort 1 so the dose was never de-escalated, Cohort -1 never opened to enrollment.
Arm/Group | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 3/3 | 6/6 | 5/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 6/6 | 6/6
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) (N=0) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) (N=3) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) (N=6) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab (N=6)
Sepsis (Infections and infestations) | 0 | 2 | 0 | 3 — * 1 patient in Cohort 1 also had secondary AE of GI bleed * 1 patient in Cohort 1 also had Anemia, Fever, Dyspnea, Biliary tract infection * 1 patient in Phase 2 also had fever, chills, blood bilirubin increase, abdominal pain.
Hepatobiliary disorder - Other:Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 0 — -1 patient in Cohort 2 also had secondary AE of small bowel obstruction
Fever (General disorders) | 0 | 2 | 0 | 0
GI bleed (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic Infection (Infections and infestations) | 0 | 1 | 0 | 0 — -1 patient in cohort 1 had secondary AE of fever.
Gastric outlet obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — -1 patient in cohort 1 had secondary AE of abdominal pain.
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — -1 patient in cohort 2 also had secondary AE of Anemia, lightheadedness, dizziness, hypotension.
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 — -1 patient in Cohort 2 also had Hyponatremia, Death NOS.
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Movements Involuntary (Nervous system disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1:Cohort-1 (Velaparib 200 mg PO Twice Daily + Nivolumab) (N=0) | Phase 1:Cohort 1 (Velaparib 300 mg PO Twice Daily + Nivolumab) (N=3) | Phase 1:Cohort 2 (Velaparib 400 mg PO Twice Daily + Nivolumab) (N=6) | Phase 2 MTD: Velaparib 400 mg PO Twice Daily + Nivolumab (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 2 | 5 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 5 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 2 | 3
Blurred vision (Eye disorders) | 0 | 0 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2
Creatinine increased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 5 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 2 | 2
Fatigue (General disorders) | 0 | 2 | 4 | 3
Fever (General disorders) | 0 | 2 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 2 | 3 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Colon infection (Infections and infestations) | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 2
Irritability (General disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 3 | 5 | 4
Malaise (General disorders) | 0 | 1 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 4 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 3 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Weight loss (Investigations) | 0 | 2 | 4 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 1 | 0
Melena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Esophageal varices (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Transient cholangitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Increased bowel frequency (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Leg cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The original accrual goal was 50 patients. Due to funding issues the accrual goal was reduced to 15 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT03061188/Prot_SAP_000.pdf